CLINICAL TRIAL: NCT06557239
Title: Salivary Oxytocin as a Biomarker in Psychedelic Assisted Psychotherapy for Anxiety and Depression: a Pilot Study
Brief Title: Salivary Oxytocin as a Biomarker in Psychedelic Assisted Psychotherapy
Acronym: PAP_OXT
Status: Completed | Type: Observational
Sponsor: Tatiana Aboulafia Brakha (Other)
Responsible Party: Sponsor-Investigator, Tatiana Aboulafia Brakha, Principal Investigator-Head of psychologists, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Other Study IDs: 2024-01122
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-08

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva- Salivary oxytocin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide (LSD) — one single dose of LSD in the context of psychedelic assisted psychotherapy as a part of a clinical routine in our department

SUMMARY:
The main objective of this pilot study is to obtain preliminary data on the reactivity of salivary oxytocin during a single LSD intake as part of PAP treatment for anxiety disorders or depression (treatment authorisations granted in advance by the Federal Officie of Public Health for compassionate use of the substance).

There will be no interference with the usual clinical routine in our Service. The protocol is only for taking additional saliva measurements to measure oxytocin levels on the day of treatment.

Participants will be asked to give 4 saliva samples the day of their LSD treatment .In addition they will fill-in self-report questionnaires which are part of the clinical routine

ELIGIBILITY:
Inclusion Criteria:

* ongoing psychotherapy with a certified psychotherapist, anxiety disorder or depression resistant to usual treatments, agreement to stop necessary medication

Exclusion Criteria:

* Exclusion: psychotic or bipolar disorder, high suicidal risk, severe cardiovascular disease, severe liver disease, neurological disease of the central nervous system, pregnancy and breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be selected from consecutive patients in the Addiction Department who have received approval from the Federal office of Public healthfor compassionate treatment with LSD as part of Psychedelic assisted psychotherapy for refractory anxiety disorder or depression. ol. Main criteria: Inclusion:
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Salivary oxytocin | the day of treatment administration (one day)
  oxytocin sampled in the saliva

SECONDARY OUTCOMES:
Self-reported symptoms of anxiety (STAI-T) | over 6 months
  State-Trait Anxiety Inventory (trait), total scores ranging from 20 to 80, higher scores indicating higher anxiety
Self-reported depressive symptoms (BDI-II) | over 6 months
  Beck Depresion Inventory-II, total scores ranging from 0 to 63, higher scores indicating higher depressive symptoms
Self-reported intensity of mystical experience | The 1 day of treatment administration
  Assessed with the self-report Mystical experience Questionnaire (MEQ-30) with total man score ranging from 0 to 5, with higher scores indicating higher intensity of mystical experience
Self-reported intensity of Connectedness | The 1 day of treatment administration
  Assessed with the self-report Watts Connectedness Scale,total mean score ranging from 0 to 100, with higher scores indicating higher connectedess

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided